CLINICAL TRIAL: NCT06010836
Title: Anesthesiology Counseling, Consent, & Professionalism
Brief Title: Anesthesia Counseling, Consent, & Professionalism
Acronym: ACCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00268333
Record Dates: First submitted 2023-05-29; First posted 2023-08-25 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Communication; Preoperative; Ethics
Keywords: Communication; Medical ethics; Professionalism
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Group getting standard treatment without script guided intervention in the preoperative period
- Script guided intervention (Experimental): Group getting script guided intervention during the preoperative conversation
  Interventions: Behavioral: Script guided conversation

INTERVENTIONS:
Behavioral: Script guided conversation — Patients getting script guided intervention of 3 domains in the preoperative period
  Arms: Script guided intervention

SUMMARY:
The anesthesia consent form has become a standard before surgery. However, verbal aspects of anesthesia consent and of the value of the preoperative anesthesia discussion has not been addressed. This study will use preoperative discussions and postoperative patient questionnaires to examine the degree of awareness that the patients and the patients families have regarding what general anesthesia is, the responsibilities of the anesthesiologist, and the specifics of what the participants are agreeing to by signing the consent form.

DETAILED DESCRIPTION:
There is a substantial body of work regarding the written anesthesia consent form. As a result, the written anesthesia consent form has become a standard requirement throughout the United States of America. However, there has been little examination of verbal aspects of anesthesia consent and of the value of the preoperative anesthesia discussion that should take place prior to surgery. Non-anesthesia medical studies have indicated that inadequate patient-physician communication and an inadequate patient-physician relationship will result in misunderstanding and an increased malpractice risk. Lack of understanding of the duties and responsibilities of anesthesiologists is also damaging to the professional status of the field of anesthesiology. This study will utilize patient interviews and questionnaires to examine the degree of awareness that the patients and the patients families possess regarding what general anesthesia is, the duties and responsibilities of the anesthesiologist, the role of the anesthesiologist within the operating room and the specifics of what the participants are agreeing to by signing the consent form. If it is determined that a more structured and thorough pre-anesthesia discussion will help patients and the patients families understand what general anesthesia is, understand the specific responsibilities of anesthesiology providers, understand the professional status of anesthesiologists, give the participants a better feeling of autonomy and better understand what the participants are agreeing to by signing the consent form, then there will be substantial ramifications to the priority and importance given to pre-anesthesia discussions nationwide. Secondary benefits include influences on anesthesia residency training and improved patient satisfaction with the anesthesia experience.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and up
* Elective Procedures
* English-speaking
* Consenting for general anesthesia

Exclusion Criteria:

* Obstetric patients
* Prisoners
* Emergency cases
* Patients under age 18
* Patients don't speak English
* Not consented for general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Sampson, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
None to be shared

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Script Guided Intervention
Started | 132 | 125
Completed | 121 | 113
Not Completed | 11 | 12
Not completed — Lost to Follow-up | 2 | 2
Not completed — Case cancelled by surgeon, or reoperation after surgical complication | 8 | 2
Not completed — Poor or absent audio recording for data collection | 1 | 4
Not completed — Did not receive intervention discussion | 0 | 4

BASELINE CHARACTERISTICS:
Population: Reporting data for study completers. 234 participants completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Script Guided Intervention | Total
Number analyzed (Participants) | 121 | 113 | 234
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 87 | 85 | 172
  >=65 years | 34 | 28 | 62
Age, Continuous [Mean (Full Range); unit: years] | 58 [19 to 84] | 57 [19 to 89] | 57.5 [19 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 57 | 135
  Male | 43 | 56 | 99
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 82 | 77 | 159
  Black | 30 | 25 | 55
  Hispanic | 3 | 5 | 8
  Asian | 4 | 5 | 9
  Other | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 121 | 113 | 234

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Recall Anesthesia Team Members
Description: Postoperative recall of anesthesia conversation. Recall of team members score 0-100 with higher score indicating better recall of anesthesia team members.
Time Frame: up to 3 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Script Guided Intervention
Number analyzed (Participants) | 121 | 113
Participants | 30 | 49

2. Primary Outcome: Number of Participants Who Recall Anesthetic Risks
Description: anesthesia risks, (0) don't remember any risks - (3) remembered 3 or more correctly
Time Frame: up to 3 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Script Guided Intervention
Number analyzed (Participants) | 121 | 113
Participants
  Recall 1 risk | 29 | 34
  Recall 2 risks | 22 | 36
  Recall 3 or more risks | 20 | 24
  No recall | 49 | 19
  Unknown | 1 | 0

3. Primary Outcome: Postoperative Understanding of Anesthetic Plan as Assessed by the Questionnaire Developed by the Study Team
Description: Demonstrate understanding of anesthetic plan; score total 0-100 with a higher score more understanding. Standard deviation is reported.
Time Frame: up to 3 days after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Script Guided Intervention
Number analyzed (Participants) | 121 | 113
score on a scale | 0.16 (0.305) | 0.714 (0.428)

4. Secondary Outcome: Number of Participants Satisfied With Anesthesia Conversation
Description: Number of participants satisfied with anesthetic conversation assessed by questionnaire developed by study team; using likert scale rating; extremely satisfied (5) to extremely dissatisfied (1)
Time Frame: up to three days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Script Guided Intervention
Number analyzed (Participants) | 121 | 113
Participants
  Satisfied | 118 | 113
  Neutral | 3 | 0
  Not satisfied | 0 | 0

5. Secondary Outcome: Preoperative Anxiety as Assessed by Questionnaire Developed by Study Team
Description: Patients are asked about any change in anxiety after the preoperative conversation using likert scale extremely reduced (5) to extremely more anxious (1)
Time Frame: up to 3 days after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Script Guided Intervention
Number analyzed (Participants) | 121 | 113
score on a scale | 3.33 (0.793) | 3.70 (0.938)

ADVERSE EVENTS:
Description: Adverse Events were not collected
Arm/Group | Control | Script Guided Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT06010836/Prot_SAP_000.pdf